CLINICAL TRIAL: NCT07248176
Title: A Clinical Study on the Safety and Efficacy of Allogeneic CAR T Cells Targeting BCMA in the Treatment of Adult r/r Multiple Myeloma
Brief Title: Universal CAR-T Cell Therapy for MM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bioray Laboratories (Industry)
Collaborators: Shanghai Tongji Hospital (Tongji Hospital of Tongji University) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-BRL-305-01-IIT
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 5.0-10×10^6cells/kg
  Interventions: Drug: Targeted BCMA Gene-Modified Allogeneic Chimeric Antigen Receptor T-Cell Injection

INTERVENTIONS:
Drug: Targeted BCMA Gene-Modified Allogeneic Chimeric Antigen Receptor T-Cell Injection — The study drug is administered intravenously at a fixed dose within 1-2 days after lymphocyte depletion, and its efficacy and safety are observed.
  Other Names: BRL-305

SUMMARY:
This trial aims to evaluate the safety and efficacy of BCMA-UCART in treating patients with r/r multiple myeloma.

DETAILED DESCRIPTION:
This study is a non-randomized, open-label, single-arm clinical trial designed to assess the efficacy and safety of combination therapy for r/r multiple myeloma using universal CAR-T cells targeting BCMA .

ELIGIBILITY:
Inclusion Criteria:

1. Expected survival of at least 3 months;
2. Subjects should have measurable disease that meets the IMWG 2016 criteria;
3. Previously received at least two lines of prior anti-myeloma therapy ；
4. Relapse , failure to achieve at least a minimal response, or disease progression after the last treatment ；
5. BCMA positive；
6. ECOG score 0-1；
7. No severe impairment or suppression of liver, kidney, coagulation, bone marrow, or lung function.

Exclusion Criteria:

1. Pregnant or breastfeeding women;
2. History of other malignant tumors;
3. Active autoimmune diseases requiring immunotherapy;
4. Previously received allogeneic stem cell transplantation;
5. Previous use of CAR-T cells or other genetically modified T cell therapies;
6. Previously received targeted BCMA therapy;
7. Severe cardiovascular disease;
8. Active infection;
9. Positive virology test;
10. Clinically significant central nervous system (CNS) diseases or pathological changes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2028-04-18 (Estimated)

PRIMARY OUTCOMES:
DLT | Within 28 Days After BRL-305 Infusion
  The number and severity of dose-limiting toxicity (DLT) events
AEs | Up to 24 Months After BRL-305 Infusion
  The total number, incidence, and severity of AEs

CONTACTS AND LOCATIONS:
Overall Officials: Ping Li, PhD, Study Director — 13564181131
Locations (1):
- Shanghi Tongji Hospital (Tongji Hospital of Tongji University), Shanghai, China

IPD SHARING:
Plan to Share IPD: No